CLINICAL TRIAL: NCT05224752
Title: Workplace Violence, Hostility & Safety
Status: Withdrawn | Type: Observational
Why Stopped: The study was merged with a different study.
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 027.NUR.2021.R
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2022-12

CONDITIONS: Violence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthcare workers at MRMC: healthcare workers at MRMC
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Online survey void of individual traceable identifiers, and launched via the Survey Monkey® portal

SUMMARY:
Workplace violence has been documented as a global, epidemic healthcare- related problem. The American Nurses Association (ANA) describes customer/client violence as an assault from a member of the public with whom the nurse interacts during the course of their regular duties. According to the ANA's website, types of violence that contribute to unsafe work environments are varying. However the customer/client violence type is prevalently experienced in healthcare, and 1 in 4 nurses are abused and experience workplace violence.

DETAILED DESCRIPTION:
Based on anecdotal reports at MRMC, and as a follow up to a 2020 research study, evidence-based practice research council (EBPRC) members and staff asked colleagues about stress-producing events in their scope of work. It was reported that individuals were unclear about available resources and preparation to handle unsafe environments when client/visitor behaviors escalated to aggressive or unsafe situations. The EBPRC members reviewed the MRMC policies related to violence/assault/injury towards MRMC personnel. What remains unclear is if staff are aware of existing policies and are adhering to reporting guidelines pertaining to employee and stakeholder safety. Additionally, based on literature review, the problem of workplace violence perpetrated by patients and visitors is excessive and escalating nationally and internationally. Additionally, at MRMC, the EBPRC acquired documentation of the number of reported assaults, aggressive behavior or violence of stakeholders (patients and visitors) towards healthcare providers that were documented and referred to the MRMC employee health services. From the local hospital's tally, there were 28 cases from January, 10, 2020 to February 4, 2021. Of the 28 cases, seven occurred between February 2, 2021 and February 4, 2021. Hence, it is essential to conduct a study targeting healthcare workers at MRMC to identify opportunities for further intervention that creates a safety-focused, supportive culture.

The Occupational Safety and Health Act and the Occupational Safety and Health Administration require that employees and employers work together to prevent or abate recognized hazardous and cited workplace areas for concerns and develop a successful safety and health management system especially for Healthcare and Social Services workers.

ELIGIBILITY:
Inclusion Criteria:

* must be a full-time, part-time or PRN [per diem] employee of MRMC
* who cares for or has contact with patients and visitors
* able to read and understand English

Exclusion Criteria:

* Individuals who are not full-time, part-time or PRN employees of MRMC who cares for or has contact with patient s and visitors

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: full-time, part-time or PRN [per diem] employee of MRMC, who cares for or has contact with patients and visitors.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
An investigator-developed questionnaire and demographic tool | from August, 1, 2021 to September 1, 2021
  based on feedback from members of the EBPRC as well as a relevant literature review will be used to evaluate group demographic characteristics and perceived preparedness and exposure for handling aggressive patients/visitors at MRMC
Education Level | from August, 1, 2021 to September 1, 2021
  High School diploma, College Associate, College Bachelor, masters, Doctoral, other
Status of service | from August, 1, 2021 to September 1, 2021
  Full time, part-time, per diem
Years of experience at Methodist | from August, 1, 2021 to September 1, 2021
  6 months to more than 11 years
Job status/title | from August, 1, 2021 to September 1, 2021
  RN, Tech/PCT or other
Age | from August, 1, 2021 to September 1, 2021
  Current age in years
Gender | from August, 1, 2021 to September 1, 2021
  Male or female
Ethnicity | from August, 1, 2021 to September 1, 2021
  Caucasian/white , Black/African American, Hispanic, Asian, or other
Which, if any, items do you consider an act of physical abuse or violence in the workplace | from August, 1, 2021 to September 1, 2021
  Hitting, Slapping, Biting, Spitting, Throwing or other
Have you ever experienced physical abuse at MRMC that involved a patient/visitor, within the last two years? | from August, 1, 2021 to September 1, 2021
  Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Adegbola,, PH.D., Principal Investigator — Methodist Health System
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data